CLINICAL TRIAL: NCT02341404
Title: An Open, Single Dose, Antitumour Effect Study of 2-hydroxy-flutamide as a Controlled Release Product (Liproca Depot), Injected Into the Prostate in Patients With Localized Prostate Cancer
Brief Title: A Study of 2-hydroxyflutamide (Liproca Depot), Injected Into the Prostate in Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lidds AB (Industry)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPC-003
Record Dates: First submitted 2014-10-17; First posted 2015-01-19 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — hydroxyflutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liproca Depot (Experimental): A parenteral controlled release depot formulation of 2-hydroxyflutamide (2-HOF) is given as a single dose injection into the prostate gland within the lobe area where the tumour tissue is localized.
  Interventions: Drug: 2-hydroxyflutamide (2-HOF)

INTERVENTIONS:
Drug: 2-hydroxyflutamide (2-HOF) — Two components are mixed, transferred to a syringe and administered with injection into the prostate
  Other Names: Liproca Depot

SUMMARY:
The primary aim of the study was to characterize and quantify the histopathological changes in the surgical specimens obtained in patients undergoing prostatectomy in addition to imaging changes (MRI) following a single injection of Liproca Depot in patients with localized prostate cancer.

DETAILED DESCRIPTION:
The primary aim of the study was to characterize and quantify the histopathological changes in the surgical specimens obtained in patients undergoing prostatectomy in addition to imaging changes (MRI) following a single injection of Liproca Depot in patients with localized prostate cancer.

The secondary aims ere to evaluate efficacy and safety of a single injection of Liproca Depot, and to follow the pharmacokinetic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years, ≤ 75 years
2. Histologically confirmed localized (stage T1c, T2a-T2c) prostate cancer that is judged relevant for prostatectomy.
3. PSA value < 20 ng/ml within 6 weeks before enrolment.
4. Gleason score ≤ 3+4 at diagnostic biopsy (or preferably with more precise method for judging the localization of the primary tumour focus (foci).
5. Adequate renal function: Creatinine < 1.5 times upper limit of normal.
6. Adequate hepatic function: Aspartate Transaminase (ASAT), Alanine Transaminase (ALAT) and Alkalase Phosphatase (ALP) < 1.5 times upper limit of normal.
7. Negative dipstick for bacteriuria.
8. Patient must have ability to cope with the study procedures and to return to scheduled visits including follow up visit.
9. Patients that has been scheduled for prostatectomy

Exclusion Criteria:

1. Ongoing or previous hormone therapy for prostate cancer.
2. On-going or previous therapy within 12 month of finasteride or dutasteride.
3. On-going or previous invasive therapy for benign prostate hyperplasia (TURP, TUMT).
4. Use of pace maker or other electronic devices
5. Symptoms or signs of acute prostatitis.
6. Symptoms or signs of ulcered proctitis
7. Severe micturation symptoms
8. On-going therapy with anticoagulant (e.g Warfarin. Other anticoagulant should be withdrawn 1 week before injection).
9. Concomitant systemic treatment with corticosteroids, or immune modulating agents.
10. Known immunosuppressive disease (e.g. HIV, diabetes).
11. Simultaneous participation in any other study involving not market authorized drugs or having participated in a study within the last 12 months prior to start of study treatment.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Characterization and quantification of histopathological measurement of tumour tissue obtained from diagnostic biopsy. | Day 1
Characterization and quantification of histopathological measurement of tumour tissue in surgical specimens obtained from patients undergoing prostatectomy | Six weeks
The diffusion/flow of tissue water (ADC) before and after treatment assessed by diffusion-weighted imaging (MRI) | Six weeks

SECONDARY OUTCOMES:
Concentration of Choline, Creatinine and Citrate in tumour tissue before and after treatment | Six weeks
Surface fraction and volume of treated tumour focus (foci) based on MRI and histopathological map from surgical specimens at baseline and end of study, respectively | Six weeks
Concentration of Plasma Prostate Specific Antigen (PSA) | Six weeks
Total prostate volume by histopathology/MRI measúrements | Six weeks
Number of participants with Adverse Events as a measure of Safety and Tolerability | Six weeks
Number of abnormal, clinically relevant, parameters from laboratory analyses | Six weeks
Pharmacokinetics (Tmax and Cmax) of 2-hydroxyflutamide (2-HOF) | Six weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Dept of Urology, University Hospital, Tampere, Finland
- Dept of Urology, University Hospital, Uppsala, Uppsala County, Sweden